CLINICAL TRIAL: NCT05139732
Title: Exploring Functional Paralysis with Advanced Magnetic Resonance Modalities
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2021-10
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-03

CONDITIONS: Functional Neurological Symptom Disorder; Paralysis; Conversion Disorder with Weakness/Paralysis
MeSH Terms: conditions — Conversion Disorder; Paralysis | interventions — Magnetic Resonance Imaging; Diffusion Tensor Imaging; Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- control: Healthy participants
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Functional Neurological Disorder (FND): People with the subtype functional paralysis
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Spinal Cord Injury (SCI): Incomplete and complete paralysis with the ability to hold a pen
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — In order to investigate the metabolic profile, magnetic resonance spectroscopy (MRS) will be applied. Functional MRI (fMRI) allows to indirectly track cell activation measuring the blood-level dependent signal changes followed spontaneously (in resting state) or evoked by a task. Diffusion weighted imaging (DWI) is based on the differences in motion of the water molecules given by the underlying microarchitecture of the nervous tissue. Diffusion tensor imaging (DTI) allows visualisation of the nerve bundles and alterations thereof. Thus, microstructural alterations can be measured.
  Other Names: Functional Magnetic Resonance Imaging (fMRI); In-vivo Magnetic Resonance Spectroscopy (MRS); Diffusion Tensor Imaging (DTI); Diffusion Weighted Imaging (DWI)

SUMMARY:
In functional neurological disorder (FND), neurological symptoms are present, such as paralysis, weakness and disturbed sensation of limbs, although clinically no abnormalities can be found. It is a poorly understood disorder with uncertain diagnosis, treatment and prognosis. In this study, the subtype functional paralysis is investigated with advanced neuroimaging techniques that go beyond standard clinical examinations. In previous research on FND, healthy volunteers have generally been used as a control group. However, since people with functional paralysis have similar symptoms to people with spinal cord injuries (SCI), it is intended to compare the three groups to find similarities and differences. With the proposed methods, the goal is to gain a detailed understanding of FND regarding nerve cell metabolism, diffusion pathways and neuronal networks involved in cognitive processes such as motor inhibition (reaction or no reaction depending on situation). Neurophysiological data, clinical assessments and questionnaires are carried out in addition to Magnetic Resonance Imaging (MRI).

The aim is to enrol 75 participants in this study, i.e. 25 people with FND, 25 people with SCI and 25 healthy control subjects.

The overall goal of the study is to find markers for FND for use in future studies to improve diagnosis and individualise therapy recommendation for both people with SCI and people with FND. Therefore, this study is a relevant step to understand FND and to diagnose this specific disease using objective MRI based diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65

Exclusion Criteria:

* Contraindication for magnetic resonance examinations (e.g. cardiac pacemaker, pregnancy, etc.)
* history of mental or neurological illness (addiction, central nervous system tumour and severe craniocerebral trauma)
* unable to hold a pen due to paralysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: FND patients are recruited at the Swiss Paraplegic Centre and the Inselspital Bern. Inpatient and outpatient SCI subjects are recruited in the Swiss Paraplegic Centre .
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Nerve Cell Metabolism | day 1
  With MRS metabolites are examined specific for cell integrity (N-acetyl-aspartate), cell energy (creatine, lactate), and neurotransmitter (choline, glutamate and glutamine).
Brain Functional Connectivity | day 1
  With fMRI in rest and task condition, the functional connectivity (FC) is examined. With that the functionally integrated relationship between spatially separated brain regions are investigated.
Fiber tracts in three dimensional mapping | day 1
  DWI provides quantitative evaluations by measuring the apparent diffusion coefficient (ADC) and fractional anisotropy (FA), which are scalars of isotropic and anisotropic diffusion. Diffusion tensor imaging (DTI) analyses the three-dimensional shape of the diffusion, also known as diffusion tensor. So, it is used to characterize the magnitude, the degree of anisotropy, and the orientation of directional diffusion of white matter.

SECONDARY OUTCOMES:
Satisfaction with Life Scale questionnaire | day 1
  Likert Scale of 1 (strong disagreement) -7 (strong agreement); 5 Questions in total
Hospital Anxiety and Depression Scale questionnaire | day 1
  Likert Scale of 1 (strong disagreement) -4 (strong agreement); 14 Questions in total
Numerical Rating Scale (NRS) questionnaire | day 1
  Rating the pain on a likert scale of 0 (no pain) -10 (insupportable pain)
Sensibility testing according to International Standards for Neurological Classification of SCI (ISNCSCI) | day 1
  A key point in each of the 28 dermatomes is tested bilaterally using light touch and pin-prick (sharp-dull discrimination). A three-point scale is used for scoring:
  0 = absent
  1. = altered (impaired or partial appreciation, including hyperesthesia)
  2. = normal or intact (similar as on the cheek) not testable

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No